CLINICAL TRIAL: NCT06052839
Title: Phase II Trial of Pulsed Dose Chemotherapy Plus Pembrolizumab in the First Line Treatment of Recurrent/Metastatic HNSCC
Brief Title: Pulsed Dose Chemotherapy Plus Pembrolizumab in Recurrent/Metastatic HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dan Zandberg (Other)
Responsible Party: Sponsor-Investigator, Dan Zandberg, Associate Professor of Medicine / Medical oncologist/hematologist, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 23-071
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma (R/M HNSCC)
Keywords: CD8 tumor infiltrating lymphocyte (TIL); interferon gamma (IFNγ); anti-PD-1 mAb
MeSH Terms: conditions — Recurrence | interventions — pembrolizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab + Carboplatin with Paclitaxel (Experimental): Pembrolizumab: Administer 200 mg intravenously (IV) every 3 weeks (q3w); maintenance will be continued at 400 mg IV q6w for 12 cycles for a total of 2 years of therapy
  Carboplatin: Started with cycle 2 (C2) of pembrolizumab and continued thereafter every 3rd cycle of pembrolizumab for a total of 4 cycles with paclitaxel; carboplatin will be given at C2, C5, C8, and C11 of pembrolizumab.
  Paclitaxel: Started with cycle 2 (C2) of pembrolizumab and continued thereafter every 3rd cycle of pembrolizumab for a total of 4 cycles with carboplatin.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Immunotherapy that works by helping the immune system to kill cancer cells by targeting and blocking a protein called PD-1 on the surface of certain immune cells called T-cells. Blocking PD-1 triggers the T-cells to find and kill cancer cells.
  Other Names: Keytruda®
Drug: Carboplatin — A chemotherapy drug that contains the metal platinum. It stops or slows the growth of cancer cells and other rapidly growing cells by damaging their DNA.
Drug: Paclitaxel — A chemotherapeutic agent used as a treatment for various cancers; paclitaxel is a mitotic inhibitor.
  Other Names: Taxol

SUMMARY:
The rationale for the new sequence of pulsed dose chemotherapy proposed in this trial is based on the hypotheses that current standard dosing of chemotherapy plus pembrolizumab ultimately suppresses the immune system and has a negative effect on the efficacy of the anti-PD-1 monoclonal antibody (mAb) therapy and that chemotherapy given after anti-PD-1 mAb therapy is associated with higher efficacy.

DETAILED DESCRIPTION:
Chemotherapy plus pembrolizumab plays a significant role in standard of care frontline treatment in R/M HNSCC and there is a need for improvement in outcomes with this combination therapy. This trial importantly will test a new dosing and sequence of pembrolizumab and chemotherapy, with the primary goal of improving efficacy but secondarily also has the potential to be better tolerated than standard dosing. Additionally, this trial may have applicability to other solid tumor types where chemotherapy and anti-PD-1 mAb are currently combined. Based on current data showing that current repetitive frequent dosing of chemotherapy may lead to immunosuppression and a detrimental effect on the prolonged duration of response expected from pembrolizumab, and that chemotherapy efficacy may be higher after anti-PD-1 mAb therapy, this trial will test a new sequence starting with pembrolizumab with less frequent dosing of chemotherapy (pulsed dose) to maximize synergy and improve efficacy. Specifically, patients will be treated with pembrolizumab 200 mg IV q3w with carboplatin/paclitaxel given starting with cycle 2 of pembrolizumab and continued thereafter every 3rd cycle of pembrolizumab (q9w) for a total of 4 cycles of carboplatin/paclitaxel. After completion of the 4th cycle of carboplatin/paclitaxel, pembrolizumab maintenance will be continued at 400 mg IV q6w for 12 cycles for a total of 2 years of therapy. Carboplatin/paclitaxel is being used as the chemotherapy doublet in this trial because there is more data for immunogenicity and higher efficacy post anti-PD-1 with taxanes, the potential to be better tolerated than infusional 5-fluorouracil (5FU), and physician preference for this chemotherapy backbone including in our Hillman network. Importantly, prior to the immunotherapy era, a phase III trial compared platinum/taxane to platinum/5FU in R/M HNSCC and found no difference in efficacy between these regimens, and outcomes in combination with pembrolizumab are comparable.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent/metastatic squamous cell carcinoma of the head and neck that is considered incurable by local therapies.
2. PD-L1 Combined Positive Score (CPS) >1
3. Age > 18 years.
4. Eastern Cooperative Oncology Group (ECOG) Performance Scale (PS) 0-2
5. Measurable disease using Response Evaluation Criteria in Solid Tumors (RECIST) 1
6. Patients must have normal organ and marrow function as defined below:

   1. absolute neutrophil count ≥1,000/mcL
   2. platelets ≥100,000/mcL
   3. total bilirubin ≤ 1.5 X the institutional upper limit of normal (ULN)
   4. AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN (≤ 5 X the institutional ULN for patients with liver metastasis)
   5. Creatinine clearance ≥40 mL/min/1.73 m2 for patients with a creatinine levels above institutional normal.
7. Female subjects of childbearing potential should have a negative urine or serum pregnancy during the screening period and also prior to receiving the first dose of study medication. If a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential should be willing to use one methods of birth control or abstain from heterosexual activity for the course of the study through 60 days after the last dose of study medication. Women of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 60 days after the last dose of study therapy.
10. Ability to understand and the willingness to sign a written informed consent document.
11. If known to have prior brain metastases, must not have evidence of active (enlarging and/or symptomatic lesions) brain disease on MRI/CT evaluation done within 30 days of consent.

Exclusion Criteria:

1. Patients should not have had prior systemic therapy alone administered in the recurrent/ or metastatic setting. If a patient received platinum based systemic therapy which was completed more than 6 months prior to signing consent given as part of multimodal curative intent treatment for locally advanced HNSCC (This includes both definitive concurrent chemoradiation and adjuvant chemoradiation) the patient is still eligible,
2. A patient cannot have received prior anti-PD-1 or anti-PD-L1 monoclonal antibody (mAb) therapy as systemic therapy for the treatment of recurrent/metastatic disease. Patients that received anti-PD-1 or anti-PD-L1 mAb therapy as part of multimodality curative intent treatment of locally advanced disease are still eligible as long as it has been at least 1 year since prior therapy. Patients that received anti-PD-1 or anti-PD-L1 mAb therapy as part of radiation for locoregional recurrence will be eligible as long as it has been 1 year since prior therapy.
3. Squamous cell carcinoma of the skin or of salivary gland origin.
4. Has an active autoimmune disease requiring systemic treatment within the past 3 months, or a syndrome that requires ongoing systemic steroids or immunosuppressive agents. Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic therapy or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism or Sjogren's syndrome will not be excluded from the study.
5. Has a history of non-infectious pneumonitis that required steroids, evidence of interstitial lung disease, or currently active non-infectious pneumonitis.
6. Prior malignancy within 2 years that in the investigator's opinion would be likely to affect the outcomes of the patients R/M HNSCC.
7. Peripheral sensory neuropathy > grade 2 by CTCAE v5.0
8. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
9. Known allergy or hypersensitivity to carboplatin, other platinum agents, pembrolizumab, or paclitaxel.
10. Baseline neutrophil count of < 1,500 cells/mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month Progression-free Survival (PFS) | At 6 months
  Proportion of patients alive and without disease progression at 6 months after starting treatment, per RECIST v1.1. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).

SECONDARY OUTCOMES:
Adverse Events (AE) and Serious Adverse Events (SAE) Related to Treatment | Up to 2 years
  Proportion of patients that experience Adverse Events or Serious Adverse Events related to treatment, per CTCAE v5.0. The maximum grade for each toxicity type will be recorded for each patient.
Overall Response Rate (ORR) | Up to 2 years
  Proportion of patients with Complete Response (CR) or Partial Response (PR) per RECIST v1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Duration of Response (DOR) | Up to 4 years
  Time from start of treatment to disease progression or death in patients who achieve Complete Response (CR) or Partial Response (PR) per RECIST v1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Overall Survival (OS) | Up to 4 years
  Median number of months from start of treatment that patients remain alive.

CONTACTS AND LOCATIONS:
Overall Officials: Dan P Zandberg, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No